CLINICAL TRIAL: NCT03994965
Title: Identification of a Serotonin 2A Receptor Subtype of Schizophrenia Spectrum Disorders With Pimavanserin: The Sub-Sero Proof-of-principle Study
Brief Title: The Sub-Sero Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug supply withdrawn (dec 2019)
Sponsor: Bjorn H. Ebdrup (Other)
Collaborators: Rigshospitalet, Denmark (Other); GCP unit, Copenhagen University Hospital (Unknown); ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor-Investigator, Bjorn H. Ebdrup, MD PhD, associate professor, vice-chair of research CNSR, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-001722-10
Record Dates: First submitted 2019-06-05; First posted 2019-06-21 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia; Psychosis
Keywords: Pimavanserin; serotonin 2AR; MR; PET
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — pimavanserin

STUDY DESIGN:
Intervention Model Description: Proof-of-principle study, investigator initiated, open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients (Experimental): 40 antipsychotic-free, first-episode schizophrenia spectrum patients will receive 6 weeks of treatment with a selective serotonin 2A Receptor (2AR) blockade.
  Before initiation of treatment patients will undergo: positron emission tomography (PET) imaging of the serotonin 2AR binding potential using the radioligand [¹¹C]Cimbi-36; magnetic resonance spectroscopy (MRS) of cerebral glutamate levels; structural Magnetic Resonance Imaging (MRI), including diffusion tensor imaging (DTI); cognitive and psychopathological examinations; Electrocardiography (ECG), and blood sampling for genetic- and metabolic analyses.
  (Full description will be updated on approval).
  Interventions: Drug: Pimavanserin 34 milligrams (MG) [Nuplazid]

INTERVENTIONS:
Drug: Pimavanserin 34 milligrams (MG) [Nuplazid] — Daily treatment with 34 mg per os for 6 weeks. Followed by a wash-out period up to 14 days, do to the theoretical risk of corrected QT interval (QTc) prolongation. Conventional anti-psychotic treatment will be initiated only upon normal ECG.

SUMMARY:
Schizophrenia is a severe, often chronic mental disorder, characterized by positive and negative symptoms and cognitive deficits. The serotonin hypothesis of schizophrenia was proposed in the 1950s, but only recently, pimavanserin, the first antipsychotic medication with selective affinity for the serotonin 2A receptor was approved.

The aim of this translational proposal is to test the clinical validity of the serotonin hypothesis of schizophrenia and to guide development of operational, objective criteria for stratification of first-episode schizophrenia spectrum patients before antipsychotic treatment.

Our previous data have strongly suggested, that a subgroup of antipsychotic-naïve patients will respond to serotonin 2A receptor (2AR) blockade. This treatment will cause minimal side-effects compared with conventional dopamine D2/3 receptor blockade.

In this Danish, investigator-initiated trial, we will establish a cohort of 40 antipsychotic-free, first-episode schizophrenia spectrum patients and enrol them in a 6-week open label, one-armed trial with selective serotonin 2AR blockade (pimavanserin).

Before initiation of pimavanserin patients will undergo: positron emission tomography (PET) imaging of the serotonin 2AR binding potential using the radioligand [¹¹C]Cimbi-36; magnetic resonance spectroscopy (MRS) of cerebral glutamate levels; structural Magnetic Resonance imaging (MRI), including Diffusion Tensor Imaging (DTI); cognitive and psychopathological examinations; Electrocardiography (ECG), and blood sampling for genetic- and metabolic analyses.

Matched healthy controls will undergo parallel examinations, but not medical treatment and PET .

ACADIA Pharmaceuticals Inc. provides the study medication (pimavanserin). ACADIA had no influence on study design and will not take part in data processing or publication of the results of the study.

DETAILED DESCRIPTION:
(More information will follow on study approval).

ELIGIBILITY:
Patients - Inclusion Criteria:

* Antipsychotic-free (as defined under Exclusion Criteria below)
* Fulfilling the diagnostic criteria of schizophrenia, persistent delusional disorder, acute and transient psychotic disorders, schizoaffective disorder, other non-organic psychotic disorders and unspecified non-organic disorders (ICD-10: F20.x; F22.x; F23.x; F24.x; F25.x; F28; F29); verified by The Schedules for Clinical Assessment in Neuropsychiatry (SCAN) 2.0 interview (Wing et al. 1990)
* Age: 18-45 years
* Legally competent (In Danish: 'myndige og habile i retslig forstand')

Patients - Exclusion Criteria:

* Prior use of antipsychotic medication longer than an episode of two weeks in the previous year and/or 6 weeks lifetime, and/or antipsychotic treatment within 30 days prior to inclusion.
* Current substance abuse ICD-10 (F1x.2) or substance abuse in any period up to 3 months prior to referral (exception: tobacco/nicotine, F17.2)
* Head injury with more than 5 minutes of unconsciousness
* Any coercive measure
* Metal implanted by operation
* Pacemaker
* Pregnancy (assessed by urine human chorionic gonadotropin (HCG))
* Female patients: Unwillingness to use safe contraception (Intra Uterine Device/System or hormonal contraceptives) during the study period including the wash out period.
* Severe physical illness
* Known QT prolongation or congenital prolongation of the QT interval
* Medical history of cardiac arrhythmias, as well as other circumstances that may increase the risk of the occurrence of torsade de pointes and/or sudden death, including symptomatic bradycardia, hypokalemia or hypomagnesemia
* Current treatment with drugs known to prolong QT interval including: Class 1A antiarrhythmics (e.g., quinidine, procainamide); Class 3 antiarrhythmics (e.g., amiodarone, sotalol); certain antibiotics (e.g., gatifloxacin, moxifloxacin).
* Allergies to any of the inactive ingredients and film coat components: pregelatinized starch, magnesium stearate, microcrystalline cellulose, hypromellose, talc, titanium dioxide, polyethylene glycol, and saccharin sodium.

Healthy controls - Inclusion Criteria:

* Matched with patients on age (+/- 2 years), sex and parental socioeconomic status
* Age 18-45 years
* Legally competent (In Danish: 'myndige og habile i retslig forstand')
* Recruitment: through online advertisement (www.forsøgsperson.dk)

Healthy controls - Exclusion Criteria:

* Any psychiatric illness any first-degree relatives with known psychiatric diagnoses or physical disease
* Substance abuse during the past 3 months or positive urine-screening of illegal drugs
* Head injury with more than 5 minutes of unconsciousness
* Components of metal implanted by operation
* Pacemaker
* Pregnancy (assessed by urine HCG)
* Severe physical illness

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Reduction in positive symptoms - Clinical response in patients after 6 weeks of treatment | 6 weeks
  Reduction in the Positive and Negative Syndrome Scale (PANSS) positive subscale score [PANSS positive baseline - PANSS positive week 6].
  To assess a patient using PANSS, an approximately 45-minute clinical interview is conducted. The patient is rated from 1 to 7 on 30 different symptoms based on the interview as well as reports of family members or primary care hospital workers.[4]
  Positive scale 7 Items, (minimum score = 7, maximum score = 49)
  Negative scale 7 Items, (minimum score = 7, maximum score = 49)
  General Psychopathology scale 16 Items, (minimum score = 16, maximum score = 112)
  For the primary outcome only the chance in PANSS positive scores will be reported.

SECONDARY OUTCOMES:
Reduction in positive symptoms after week 2 and 4 - Secondary clinical endpoints | 6 weeks
  Include reduction in PANSS positive subscale score compared to baseline by week 2 and 4, respectively.
  See description of PANSS score under primary outcome.
Reduction in negative symptoms after 6 weeks of treatment, measured with the Brief Negative Symptom Scale (BNSS). | 6 weeks
  Secondary clinical endpoints, negative symptoms
  Negative symptoms will be assessed by Brief Negative Symptom Scale (BNSS). Measures 5 domains: blunted affect, alogia, asociality, anhedonia, and avolition.
  The BNSS includes a manual, score sheet, and workbook, and has 13 items organized into 6 subscales. The manual defines the terms used in the scale, provides anchors for each item, and gives instructions for a semistructured interview, including suggested questions. The workbook extracts the suggested questions and the anchors and is designed for the rater's reference during administration. All the items in the BNSS are rated on a 7-point (0-6) scale, with anchor points generally ranging from the symptom's being absent (0) to severe (6).
Reduction in obsessive symptoms after 6 weeks of treatment, measured with The Brief Obsessive Compulsive Scale (BOCS). | 6 weeks
  Secondary clinical endpoints, obsessive symptoms
  Measured by The Brief Obsessive Compulsive Scale (BOCS). The BOCS consists of a 15-item Symptom Checklist including three items (hoarding, dysmorphophobia and self-harm) related to the The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) category "Obsessive-compulsive related disorders", accompanied by a single six-item Severity Scale for obsessions and compulsions combined.
  Total severity scale (questions 1-6) score range from: 0-24. Endorsement of 2 or more items in the checklist or a mean score of 1.5 or above on the severity scale suggests an Obsessive-compulsive disorder (OCD).
  Higher mean scores on the severity scale (questions 1-6) starting on page 4 indicate higher severity.
The proportion of patients achieving symptomatic remission (using the Andreasen criteria) at week 6. | 6 weeks
  Secondary clinical endpoints, patients in remission
  Andreasen criteria:
  Positive and Negative Syndrome Scale (PANSS) Items for use in Symptoms of Remission, patients must score less than or equal to 3 (mild) on these eight items.
  Name; Item nr:
  Delusions; P1 Unusual thought content; G9 Hallucinatory behavior; P3 Conceptual disorganization; P2 Mannerisms/Posturing; G5 Blunted affect; N1 Passive social withdrawal; N4 Lack of spontaneity/Flow of Conversation; N6
The serotonin 2AR binding potential in relation to treatment response | 6 weeks
  Secondary neuropsychiatric endpoints; positron emission tomography (PET)
  In-depth characterization pre-treatment measurements of patients, who respond to serotonergic 2AR blockade.
  Analysis of PET scans regarding serotonin 2AR binding potential compared with treatment response as well as characterization of differences in sub-regions.
Characterization of response in Magnetic Resonance Imaging parameters after 6 weeks of treatment. | 6 weeks
  Secondary neuropsychiatric endpoints; MR In-depth characterization pre-treatment measurements of patients, who respond to serotonergic 2AR blockade.
  Analysis of structural MR, spectroscopy of glutamate levels and diffusion tensor imaging (DTI).
Response in cognitive functioning using CANTAB after 6 weeks of treatment. | 6 weeks
  Secondary neuropsychiatric endpoints
  In-depth characterization pre-treatment measurements of patients, who respond to serotonergic 2AR blockade.
  Neuropsychology: test of cognition using CANTAB and selected paper and pencil tests.
Characterization of para-clinical parameters in patients using both genetic high-density-snip-arrays and clinical blood markers. | 6 weeks
  To exclude other clinical diseases than schizophrenia and as a safety-measure, blood-samples are taken for somatic screening including haemoglobin, hematocrit, ferritin, white blood cells, platelet count, sodium, potassium, creatinine, carbamide, albumin, C-reactive protein (CRP), HbA1c and fasting glucose, fasting lipids, thyroid stimulating hormone, alanine and aspartate amino transferase, bilirubin, lactate dehydrogenase and alkaline phosphatase.
  The genetic-blood samples will be analysed with an array designed for population based genetic studies. We will use a high-density-snip-array of approximately 1 million snips (SNP/snip: single nucleotide polymorphism). The array will be applied to the genome in full, but genome sequencing will not be performed neither of individual genes nor the full genome. The genetic data will be used to identify a genetic risk score compared to the background population.

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn H Ebdrup, MD, PhD, Principal Investigator — University of Copenhagen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Baltzersen OB, Meltzer HY, Frokjaer VG, Raghava JM, Baandrup L, Fagerlund B, Larsson HBW, Fibiger HC, Glenthoj BY, Knudsen GM, Ebdrup BH. Identification of a Serotonin 2A Receptor Subtype of Schizophrenia Spectrum Disorders With Pimavanserin: The Sub-Sero Proof-of-Concept Trial Protocol. Front Pharmacol. 2020 Apr 30;11:591. doi: 10.3389/fphar.2020.00591. eCollection 2020. PMID 32425802